CLINICAL TRIAL: NCT06676488
Title: A Randomized Crossover Trial of Bright Light Therapy in Irritable Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00138575; P30DK123704 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome (IBS); Circadian Misalignment
Keywords: Stomach; Irritable Bowel Syndrome; Circadian Misalignment
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-Timer Device (Bright Light Therapy) (Experimental): Morning bright light therapy will be administrated through a safe wearable device called a Re-timer. The Re-Timer glasses are lightweight and deliver blue-green light at 500nm, mimicking exposure to natural light. The device emits light at a higher wavelength than the UV range and has a UV filter for added safety. Subjects will be asked to wear the glasses for one hour each morning per day for 7 days a week. They will wear the device for a total of 14 days to receive the full therapeutic effect. Additionally, subjects will be asked to complete the light therapy the first hour of being awake and remain indoors while using the device. Participants will be informed that they can wear the device freely throughout their home or work environment but should avoid activities that could potentially be harmful (i.e., driving, contact sports, operating heavy machinery).
  Interventions: Device: Re-Timer glasses
- Placebo device (non Bright Light Therapy) (Placebo Comparator): Subjects will be asked to wear glasses that do not provide Bright Light Therapy for one hour each morning per day for 7 days a week as recommended by the manufacturer. They will wear the device for a total of 14 days to receive the full therapeutic effect. Additionally, subjects will be asked to complete the light therapy the first hour of being awake and remain indoors while using the device. Participants will be informed that they can wear the device freely throughout their home or work environment but should avoid activities that could potentially be harmful (i.e., driving, contact sports, operating heavy machinery).
  Interventions: Device: Placebo Device

INTERVENTIONS:
Device: Re-Timer glasses — Morning bright light therapy (BLT) will be administered through a safe wearable glasses device called a Re-Timer, purchased from the manufacturer Re-Timer.
  Arms: Re-Timer Device (Bright Light Therapy)
Device: Placebo Device — Placebo glasses not providing Bright Light Therapy
  Arms: Placebo device (non Bright Light Therapy)

SUMMARY:
The purpose of this research study is to assess whether morning bright light therapy (BLT) using a wearable device called a Re-Timer could potentially improve Irritable Bowel Syndrome (IBS) symptoms and decrease intestinal permeability (leaky gut). Morning bright light therapy will be administrated through a safe-wearable glasses device called a Re-Timer. The Re-Timer glasses are lightweight and deliver blue-green light at 500nm, mimicking exposure to natural light.

DETAILED DESCRIPTION:
The hypothesis of this study is that morning bright light therapy (BLT) using Re-Timer™ glasses in irritable bowel syndrome (IBS) patients with circadian misalignment (CM), will improve IBS symptom severity, improve circadian misalignment, decrease intestinal permeability and improve stool microbial diversity. Our overall objective is to assess the effects of morning bright light therapy on IBS symptom severity, circadian misalignment, intestinal permeability and intestinal microbiota. We propose to conduct a 6-week, single center, randomized, crossover pilot trial involving 30 subjects with active IBS symptoms (IBS-SSS >75), and circadian misalignment (CM) based on late chronotype (Munich Chronotype Questionnaire, Corrected Midpoint of Sleep > 4:00h). Subjects will be randomized to BLT or placebo with a 2-week washout between each condition. All subjects will have assessments at two timepoints: after 2 weeks of BLT, and after 2 weeks of placebo.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years old
* Irritable Bowel Syndrome based on Rome IV diagnostic criteria
* Mild to severe IBS symptom severity based on IBS-SSS greater than or equal to 75 17.
* Late chronotype based on the Munich Chronotype Questionnaire (Corrected Midpoint of Sleep > 4:00h) 18 Exclusion Criteria
* Subject that are pregnant or plan to become pregnant.
* Night shift workers or people who have crossed more than 2 time zones in the previous 4 weeks.
* Regular use of medications that affect intestinal permeability, and/or endogenous melatonin including metoclopramide, NSAIDs, beta blockers, antibiotics, psychotropic medications, hypnotics and exogenous melatonin products during 4 weeks prior to the study.
* Any major organ disease - known renal impairment, diabetes, liver disease, or significant cardiac failure (NY classification stage III/IV), inflammatory bowel disease or celiac disease per chart review and/or medical history.
* Diagnosis of narrow angle glaucoma or retinal disorders or demonstrated symptoms indicative of these diagnosis during the eligibility screening.
* Moderate to severe depression (score ≥ 21 or any endorsement of suicidal intent on the Beck Depression Inventory) 19
* Sleep apnea (score high risk in 2 or more categories of the Berlin Questionnaire) 20
* Restless leg syndrome (score ≥ 15 on the IRLS Study Group Rating Scale) 21
* Inability or unwillingness of subject to sign an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1a | 2 weeks of morning Bright Light Therapy (BLT)
  In Aim 1a, we predict 2 weeks of morning BLT in IBS subjects with CM will improve IBS-symptom severity based on the IBS Severity Scoring Scale as compared to the control (wear the Re-Timer™ glasses without light therapy).
Aim 1b | 2 weeks of morning Bright Light Therapy (BLT)
  In Aim 1b, we predict 2 weeks of morning BLT will improve circadian misalignment as accessed by wrist actigraphy (interdaily stability, intradaily variability, and relative amplitude).

SECONDARY OUTCOMES:
Aim 2 | 2 weeks of morning Bright Light Therapy (BLT)
  Aim 2, we will evaluate the impact of BLT on intestinal barrier homeostasis in IBS as measured by 2a) intestinal permeability, urinary sucralose percent excretion after oral challenge and 2b) stool microbiota diversity using 16S ribosomal RNA sequencing. We predict that BLT will decrease intestinal permeability and improve stool microbiota diversity and structure.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Green, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Background] 19. Beck AT, Steer RA, Brown G. Beck Depression Inventory-II (BDI-II). APA PsycTests. 1996.
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Roenneberg T, Wirz-Justice A, Merrow M. Life between clocks: daily temporal patterns of human chronotypes. J Biol Rhythms. 2003 Feb;18(1):80-90. doi: 10.1177/0748730402239679. PMID 12568247
- [Background] Terman M, Terman JS. Bright light therapy: side effects and benefits across the symptom spectrum. J Clin Psychiatry. 1999 Nov;60(11):799-808; quiz 809. PMID 10584776
- [Background] Pail G, Huf W, Pjrek E, Winkler D, Willeit M, Praschak-Rieder N, Kasper S. Bright-light therapy in the treatment of mood disorders. Neuropsychobiology. 2011;64(3):152-62. doi: 10.1159/000328950. Epub 2011 Jul 29. PMID 21811085
- [Background] Micic G, Lovato N, Gradisar M, Ferguson SA, Burgess HJ, Lack LC. The etiology of delayed sleep phase disorder. Sleep Med Rev. 2016 Jun;27:29-38. doi: 10.1016/j.smrv.2015.06.004. Epub 2015 Jul 3. PMID 26434674
- [Background] Butler T, Maidstone JR, Rutter KM, McLaughlin TJ, Ray WD, Gibbs EJ. The Associations of Chronotype and Shift Work With Rheumatoid Arthritis. J Biol Rhythms. 2023 Oct;38(5):510-518. doi: 10.1177/07487304231179595. Epub 2023 Jun 29. PMID 37382359
- [Background] Hashemipour S, Yazdi Z, Mahabad N. Association of Evening Chronotype with Poor Control of Type 2 Diabetes: Roles of Sleep Duration and Insomnia Level. Int J Endocrinol Metab. 2020 Aug 30;18(3):e99701. doi: 10.5812/ijem.99701. eCollection 2020 Jul. PMID 33281907
- [Background] Piche T, Barbara G, Aubert P, Bruley des Varannes S, Dainese R, Nano JL, Cremon C, Stanghellini V, De Giorgio R, Galmiche JP, Neunlist M. Impaired intestinal barrier integrity in the colon of patients with irritable bowel syndrome: involvement of soluble mediators. Gut. 2009 Feb;58(2):196-201. doi: 10.1136/gut.2007.140806. Epub 2008 Sep 29. PMID 18824556
- [Background] Hanning N, Edwinson AL, Ceuleers H, Peters SA, De Man JG, Hassett LC, De Winter BY, Grover M. Intestinal barrier dysfunction in irritable bowel syndrome: a systematic review. Therap Adv Gastroenterol. 2021 Feb 24;14:1756284821993586. doi: 10.1177/1756284821993586. eCollection 2021. PMID 33717210
- [Background] Nojkov B, Rubenstein JH, Chey WD, Hoogerwerf WA. The impact of rotating shift work on the prevalence of irritable bowel syndrome in nurses. Am J Gastroenterol. 2010 Apr;105(4):842-7. doi: 10.1038/ajg.2010.48. Epub 2010 Feb 16. PMID 20160712
- [Background] Voigt RM, Forsyth CB, Green SJ, Mutlu E, Engen P, Vitaterna MH, Turek FW, Keshavarzian A. Circadian disorganization alters intestinal microbiota. PLoS One. 2014 May 21;9(5):e97500. doi: 10.1371/journal.pone.0097500. eCollection 2014. PMID 24848969
- [Background] Codoner-Franch P, Gombert M. Circadian rhythms in the pathogenesis of gastrointestinal diseases. World J Gastroenterol. 2018 Oct 14;24(38):4297-4303. doi: 10.3748/wjg.v24.i38.4297. PMID 30344415
- [Background] Voigt RM, Forsyth CB, Keshavarzian A. Circadian rhythms: a regulator of gastrointestinal health and dysfunction. Expert Rev Gastroenterol Hepatol. 2019 May;13(5):411-424. doi: 10.1080/17474124.2019.1595588. Epub 2019 Mar 25. PMID 30874451
- [Background] Weerts ZZRM, Masclee AAM, Witteman BJM, Clemens CHM, Winkens B, Brouwers JRBJ, Frijlink HW, Muris JWM, De Wit NJ, Essers BAB, Tack J, Snijkers JTW, Bours AMH, de Ruiter-van der Ploeg AS, Jonkers DMAE, Keszthelyi D. Efficacy and Safety of Peppermint Oil in a Randomized, Double-Blind Trial of Patients With Irritable Bowel Syndrome. Gastroenterology. 2020 Jan;158(1):123-136. doi: 10.1053/j.gastro.2019.08.026. Epub 2019 Aug 27. PMID 31470006
- [Background] Black CJ, Ford AC. Global burden of irritable bowel syndrome: trends, predictions and risk factors. Nat Rev Gastroenterol Hepatol. 2020 Aug;17(8):473-486. doi: 10.1038/s41575-020-0286-8. Epub 2020 Apr 15. PMID 32296140
- [Background] Peery AF, Crockett SD, Murphy CC, Lund JL, Dellon ES, Williams JL, Jensen ET, Shaheen NJ, Barritt AS, Lieber SR, Kochar B, Barnes EL, Fan YC, Pate V, Galanko J, Baron TH, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2018. Gastroenterology. 2019 Jan;156(1):254-272.e11. doi: 10.1053/j.gastro.2018.08.063. Epub 2018 Oct 10. PMID 30315778
- [Background] Sperber AD, Dumitrascu D, Fukudo S, Gerson C, Ghoshal UC, Gwee KA, Hungin APS, Kang JY, Minhu C, Schmulson M, Bolotin A, Friger M, Freud T, Whitehead W. The global prevalence of IBS in adults remains elusive due to the heterogeneity of studies: a Rome Foundation working team literature review. Gut. 2017 Jun;66(6):1075-1082. doi: 10.1136/gutjnl-2015-311240. Epub 2016 Jan 27. PMID 26818616
- [Background] Lacy BE, Patel NK. Rome Criteria and a Diagnostic Approach to Irritable Bowel Syndrome. J Clin Med. 2017 Oct 26;6(11):99. doi: 10.3390/jcm6110099. PMID 29072609

DOCUMENTS (1):
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT06676488/ICF_000.pdf